CLINICAL TRIAL: NCT00476827
Title: A Phase II Safety and Tolerability Study of Avastin When Added to Single-agent Chemotherapy to Treat Patient With Breast Cancer Metastatic to Brain
Brief Title: A Phase II Safety and Tolerability Study of Bevacizumab When Added to Single-agent Chemotherapy to Treat Patient With Breast Cancer Metastatic to Brain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014926; AVF4124s; 9597-07-4R0 (Other: Duke IRB Legacy Number)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic; Brain; Anti-angiogenesis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Docetaxel; Irinotecan; Paclitaxel; Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Bevacizumab / Capecitabine (Active Comparator): Bevacizumab 15 mg/kg every 3 weeks in combination with Capecitabine (Xeloda), 2 weeks on and 1 week off on a every 3 week cycle.
  Interventions: Drug: Bevacizumab
- Bevacizumab / Docetaxel (Active Comparator): Docetaxel (taxotere) 35mg/m² IV over 60 min days 1, 8, and 15 in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: Docetaxel
- Bevacizumab /Irinotecan (Camptosar®, CPT-11) (Active Comparator): CPT-11 (Irinotecan, Camptosar) - Patients being treated with an enzyme inducing antiepileptic drug (EIAED) will receive 340 mg/m² IV; others will receive 125 mg/m² IV 90 min on days 1 and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: CPT-11
- Bevacizumab / Paclitaxel (Active Comparator): Paclitaxel (Taxol)90 mg/m2 IV over 60-90 min days 1, 8, and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: Paclitaxel
- Bevacizumab /Vinorelbine Tartrate (Active Comparator): Vinorelbine Tartrate (Navelbine®) 25 mg/m² IV over 10 min days 1, 8 and 15 in combination with avastin 10 mg/kg IV on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: Vinorelbine Tartrate
- Bevacizumab / Gemcitabine (Active Comparator): Gemcitabine (difluorodeoxycytidine, dFdC) 1000 mg/m2 IV on days 1 and 8 in combination with avastin 15 mg/kg IV on day 1 of a 21-day treatment cycle.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab(Avastin) 15 mg/kg every 3 weeks in combination with Capecitabine (Xeloda), 2 weeks on and 1 week off on a every 3 week cycle. until progression or unacceptable toxicity develops
  Other Names: Avastin
  Arms: Bevacizumab / Capecitabine
Drug: Docetaxel — Docetaxel 35mg/m² IV over 60 min days 1, 8, and 15 in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle. until progression or unacceptable toxicity develops
  Other Names: Taxotere
  Arms: Bevacizumab / Docetaxel
Drug: CPT-11 — CPT-11 (Irinotecan, Camptosar) - Patients being treated with an enzyme inducing antiepileptic drug (EIAED) will receive 340 mg/m² IV; others will receive 125 mg/m² IV 90 min on days 1 and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.until progression or unacceptable toxicity develops
  Other Names: Irinotecan; Camptosar
  Arms: Bevacizumab /Irinotecan (Camptosar®, CPT-11)
Drug: Paclitaxel — Paclitaxel (Taxol)90 mg/m2 IV over 60-90 min days 1, 8, and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.until progression or unacceptable toxicity develops
  Other Names: Taxol
  Arms: Bevacizumab / Paclitaxel
Drug: Vinorelbine Tartrate — Vinorelbine Tartrate (Navelbine®) 25 mg/m² IV over 10 min days 1, 8 and 15 in combination with avastin 10 mg/kg IV on days 1 and 15 of a 28-day cycle. until progression or unacceptable toxicity develops
  Other Names: Navelbine®
  Arms: Bevacizumab /Vinorelbine Tartrate
Drug: Gemcitabine — Gemcitabine (difluorodeoxycytidine, dFdC) 1000 mg/m2 IV on days 1 and 8 in combination with avastin 15 mg/kg IV on day 1 of a 21-day treatment cycle.until progression or unacceptable toxicity develops
  Other Names: difluorodeoxycytidine
  Arms: Bevacizumab / Gemcitabine

SUMMARY:
Our hypothesis is that this study design, in which bevacizumab is added to one of six single agent chemotherapies with proven activity in metastatic breast cancer, will result in regression or stabilization of this disease in a safe and tolerable manner.

DETAILED DESCRIPTION:
There is an unmet clinical need for effective therapy of breast cancer that has metastasized to the brain. In this scenario, median survival is around 12 months using currently available therapeutic interventions. The majority of chemotherapy-based clinical trials have considered the presence of central nervous system metastasis an exclusion criterion due to the risk of toxicities, the inability of chemotherapeutic agents to cross the blood brain barrier, and the limited overall survival within this patient population.

The preclinical data regarding the safety and activity of bevacizumab in vascular endothelial growth factor(VEGF)-expressing tumors provide a good rationale for its study in patients with breast cancer with metastasis to the brain. Yano, et al. illustrated that tumor cell expression of VEGF messenger ribonucleic acid and protein directly correlated with angiogenesis and growth of brain metastasis in a nude mouse model. Transfecting the experimental cell lines known to produce visceral metastasis with an anti-sense VEGF-gene significantly reduced the incidence of brain metastasis. Kim, et al. illustrated that a murine model specific for brain metastases originating from breast cancer showed elevated expression of the angiogenic and permeability-inducing factor VEGF-A. The growth of the brain metastases in this model was attenuated by the addition of a VEGF-tyrosine kinase inhibitor via induction of apoptosis and decreased angiogenesis. VEGF has also been implicated in the development of brain edema, a significant source of the morbidity and mortality associated with brain metastasis. Enhanced levels of VEGF and its receptors have been reported in a murine model after induction of cortical ischemia. Finally, antagonism of VEGF was demonstrated to reduce both immediate and delayed volume of infarct.

The optimal dose of bevacizumab has been extensively studied in phase I trials alone and in combination with chemotherapy. The safe and effective dose has been established as 10 mg/kg q 14 days or 15 mg/kg Q 21 days. In addition to irinotecan and paclitaxel, it has been previously used in phase II/III settings in combination with capecitabine, vinorelbine, gemcitabine, and docetaxel. Phase III studies showed an overall survival advantage when bevacizumab was added to an irinotecan/Fluorouracil (5FU)-based regimen for metastatic colorectal cancer, and when added to weekly paclitaxel for metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18+, with evaluable metastatic breast cancer and stable brain metastases
* Must have received definitive radiotherapy
* No evidence, or history of, central nervous system hemorrhage
* Adequate organ and hematological function

Exclusion Criteria:

* Active infection, non-healing wound, or history of any bleeding diathesis or coagulopathy
* Uncontrolled hypertension, congestive heart failure, peripheral vascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Palm Beach Cancer Center Institute, West Palm Beach, Florida
  - Presbyterian Health Care, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Virginia Oncology Associates, Newport News, Virginia

REFERENCES:
- [Background] Kirsch DG, Loeffler JS. Brain metastases in patients with breast cancer: new horizons. Clin Breast Cancer. 2005 Jun;6(2):115-24. doi: 10.3816/CBC.2005.n.013. PMID 16001989
- [Background] Boogerd W, Vos VW, Hart AA, Baris G. Brain metastases in breast cancer; natural history, prognostic factors and outcome. J Neurooncol. 1993 Feb;15(2):165-74. doi: 10.1007/BF01053937. PMID 8509821
- [Background] Lin NU, Bellon JR, Winer EP. CNS metastases in breast cancer. J Clin Oncol. 2004 Sep 1;22(17):3608-17. doi: 10.1200/JCO.2004.01.175. PMID 15337811
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Engel J, Eckel R, Aydemir U, Aydemir S, Kerr J, Schlesinger-Raab A, Dirschedl P, Holzel D. Determinants and prognoses of locoregional and distant progression in breast cancer. Int J Radiat Oncol Biol Phys. 2003 Apr 1;55(5):1186-95. doi: 10.1016/s0360-3016(02)04476-0. PMID 12654426
- [Background] Patchell RA, Tibbs PA, Walsh JW, Dempsey RJ, Maruyama Y, Kryscio RJ, Markesbery WR, Macdonald JS, Young B. A randomized trial of surgery in the treatment of single metastases to the brain. N Engl J Med. 1990 Feb 22;322(8):494-500. doi: 10.1056/NEJM199002223220802. PMID 2405271
- [Background] Lederman G, Wronski M, Fine M. Fractionated radiosurgery for brain metastases in 43 patients with breast carcinoma. Breast Cancer Res Treat. 2001 Jan;65(2):145-54. doi: 10.1023/a:1006490200335. PMID 11261830
- [Background] Firlik KS, Kondziolka D, Flickinger JC, Lunsford LD. Stereotactic radiosurgery for brain metastases from breast cancer. Ann Surg Oncol. 2000 Jun;7(5):333-8. doi: 10.1007/s10434-000-0333-1. PMID 10864339
- [Background] Folkman J. Tumor angiogenesis: therapeutic implications. N Engl J Med. 1971 Nov 18;285(21):1182-6. doi: 10.1056/NEJM197111182852108. No abstract available. PMID 4938153
- [Background] Ferrara N, Gerber HP, LeCouter J. The biology of VEGF and its receptors. Nat Med. 2003 Jun;9(6):669-76. doi: 10.1038/nm0603-669. PMID 12778165
- [Background] Takahashi Y, Kitadai Y, Bucana CD, Cleary KR, Ellis LM. Expression of vascular endothelial growth factor and its receptor, KDR, correlates with vascularity, metastasis, and proliferation of human colon cancer. Cancer Res. 1995 Sep 15;55(18):3964-8. PMID 7664263
- [Background] Brown LF, Berse B, Jackman RW, Tognazzi K, Guidi AJ, Dvorak HF, Senger DR, Connolly JL, Schnitt SJ. Expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in breast cancer. Hum Pathol. 1995 Jan;26(1):86-91. doi: 10.1016/0046-8177(95)90119-1. PMID 7821921
- [Background] Na X, Wu G, Ryan CK, Schoen SR, di'Santagnese PA, Messing EM. Overproduction of vascular endothelial growth factor related to von Hippel-Lindau tumor suppressor gene mutations and hypoxia-inducible factor-1 alpha expression in renal cell carcinomas. J Urol. 2003 Aug;170(2 Pt 1):588-92. doi: 10.1097/01.ju.0000074870.54671.98. PMID 12853836
- [Background] Fontanini G, Bigini D, Vignati S, Basolo F, Mussi A, Lucchi M, Chine S, Angeletti CA, Harris AL, Bevilacqua G. Microvessel count predicts metastatic disease and survival in non-small cell lung cancer. J Pathol. 1995 Sep;177(1):57-63. doi: 10.1002/path.1711770110. PMID 7472781
- [Background] Schneider BP, Miller KD. Angiogenesis of breast cancer. J Clin Oncol. 2005 Mar 10;23(8):1782-90. doi: 10.1200/JCO.2005.12.017. No abstract available. PMID 15755986
- [Background] Relf M, LeJeune S, Scott PA, Fox S, Smith K, Leek R, Moghaddam A, Whitehouse R, Bicknell R, Harris AL. Expression of the angiogenic factors vascular endothelial cell growth factor, acidic and basic fibroblast growth factor, tumor growth factor beta-1, platelet-derived endothelial cell growth factor, placenta growth factor, and pleiotrophin in human primary breast cancer and its relation to angiogenesis. Cancer Res. 1997 Mar 1;57(5):963-9. PMID 9041202
- [Background] Ferrara N. Role of vascular endothelial growth factor in the regulation of angiogenesis. Kidney Int. 1999 Sep;56(3):794-814. doi: 10.1046/j.1523-1755.1999.00610.x. PMID 10469350
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Miller KD, et al. E2100: a randomized phase III trial of paclitaxel vs paclitaxel plus bevacizumab as first-line therapy for locally recurrent or metastatic breast cancer. Proc: ASCO 2005; (#3) (Abstract).
- [Background] Yano S, Shinohara H, Herbst RS, Kuniyasu H, Bucana CD, Ellis LM, Davis DW, McConkey DJ, Fidler IJ. Expression of vascular endothelial growth factor is necessary but not sufficient for production and growth of brain metastasis. Cancer Res. 2000 Sep 1;60(17):4959-67. PMID 10987313
- [Background] Salmaggi A, Eoli M, Frigerio S, Silvani A, Gelati M, Corsini E, Broggi G, Boiardi A. Intracavitary VEGF, bFGF, IL-8, IL-12 levels in primary and recurrent malignant glioma. J Neurooncol. 2003 May;62(3):297-303. doi: 10.1023/a:1023367223575. PMID 12777082
- [Background] Kim LS, Huang S, Lu W, Lev DC, Price JE. Vascular endothelial growth factor expression promotes the growth of breast cancer brain metastases in nude mice. Clin Exp Metastasis. 2004;21(2):107-18. doi: 10.1023/b:clin.0000024761.00373.55. PMID 15168728
- [Background] Lamszus K, Ulbricht U, Matschke J, Brockmann MA, Fillbrandt R, Westphal M. Levels of soluble vascular endothelial growth factor (VEGF) receptor 1 in astrocytic tumors and its relation to malignancy, vascularity, and VEGF-A. Clin Cancer Res. 2003 Apr;9(4):1399-405. PMID 12684411
- [Background] Godard S, Getz G, Delorenzi M, Farmer P, Kobayashi H, Desbaillets I, Nozaki M, Diserens AC, Hamou MF, Dietrich PY, Regli L, Janzer RC, Bucher P, Stupp R, de Tribolet N, Domany E, Hegi ME. Classification of human astrocytic gliomas on the basis of gene expression: a correlated group of genes with angiogenic activity emerges as a strong predictor of subtypes. Cancer Res. 2003 Oct 15;63(20):6613-25. PMID 14583454
- [Background] Birner P, Piribauer M, Fischer I, Gatterbauer B, Marosi C, Ambros PF, Ambros IM, Bredel M, Oberhuber G, Rossler K, Budka H, Harris AL, Hainfellner JA. Vascular patterns in glioblastoma influence clinical outcome and associate with variable expression of angiogenic proteins: evidence for distinct angiogenic subtypes. Brain Pathol. 2003 Apr;13(2):133-43. doi: 10.1111/j.1750-3639.2003.tb00013.x. PMID 12744467
- [Background] Stefanik DF, Fellows WK, Rizkalla LR, Rizkalla WM, Stefanik PP, Deleo AB, Welch WC. Monoclonal antibodies to vascular endothelial growth factor (VEGF) and the VEGF receptor, FLT-1, inhibit the growth of C6 glioma in a mouse xenograft. J Neurooncol. 2001 Nov;55(2):91-100. doi: 10.1023/a:1013329832067. PMID 11817706
- [Background] Cobleigh MA, Langmuir VK, Sledge GW, Miller KD, Haney L, Novotny WF, Reimann JD, Vassel A. A phase I/II dose-escalation trial of bevacizumab in previously treated metastatic breast cancer. Semin Oncol. 2003 Oct;30(5 Suppl 16):117-24. doi: 10.1053/j.seminoncol.2003.08.013. PMID 14613032
- [Background] Vrendenburgh JJ, et al. Bevacizumab, a monoclonal antibody to VEGF, and irinotecan for the treatment of malignant gliomas. Proc: ASCO 2006;24(18S):1506.
- [Background] van Bruggen N, Thibodeaux H, Palmer JT, Lee WP, Fu L, Cairns B, Tumas D, Gerlai R, Williams SP, van Lookeren Campagne M, Ferrara N. VEGF antagonism reduces edema formation and tissue damage after ischemia/reperfusion injury in the mouse brain. J Clin Invest. 1999 Dec;104(11):1613-20. doi: 10.1172/JCI8218. PMID 10587525
- [Background] Kovacs Z, Ikezaki K, Samoto K, Inamura T, Fukui M. VEGF and flt. Expression time kinetics in rat brain infarct. Stroke. 1996 Oct;27(10):1865-72; discussion 1872-3. doi: 10.1161/01.str.27.10.1865. PMID 8841346
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Burstin HJ, et al. Phase II trial of anti-VEGF antibody bevacizumab in combination with vinorelbine for refractory advanced breast cancer. Breast Can Res Treat 2002;76(supp 1):S115.
- [Background] Kindler HL, Friberg G, Singh DA, Locker G, Nattam S, Kozloff M, Taber DA, Karrison T, Dachman A, Stadler WM, Vokes EE. Phase II trial of bevacizumab plus gemcitabine in patients with advanced pancreatic cancer. J Clin Oncol. 2005 Nov 1;23(31):8033-40. doi: 10.1200/JCO.2005.01.9661. PMID 16258101
- [Background] Ramaswamy B, Elias AD, Kelbick NT, Dodley A, Morrow M, Hauger M, Allen J, Rhoades C, Kendra K, Chen HX, Eckhardt SG, Shapiro CL. Phase II trial of bevacizumab in combination with weekly docetaxel in metastatic breast cancer patients. Clin Cancer Res. 2006 May 15;12(10):3124-9. doi: 10.1158/1078-0432.CCR-05-2603. PMID 16707611
- [Background] Genentech, Inc. Investigator's Brochure. Issued April 2006.
- [Background] Macdonald DR, Cascino TL, Schold SC Jr, Cairncross JG. Response criteria for phase II studies of supratentorial malignant glioma. J Clin Oncol. 1990 Jul;8(7):1277-80. doi: 10.1200/JCO.1990.8.7.1277. PMID 2358840
- [Background] Jung SH, Lee T, Kim K, George SL. Admissible two-stage designs for phase II cancer clinical trials. Stat Med. 2004 Feb 28;23(4):561-9. doi: 10.1002/sim.1600. PMID 14755389
- [Background] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Amer Stat Assoc 1958;43:457-81.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be identified in cancer center outpatient clinics multi-site. The study will be introduced by a physician or caregiver known to the patient. We will need to review protected health information in order to identify subjects, and information resulting from this activity will be used only to assess eligibility of a subject.
Pre-assignment Details: to meet inclusion must be 2 wks from prior hormonal chemotherapy and radio-static surgery, 4 weeks since major surgery and 8 weeks from neuro surgery. excluded for prior tx with avastin or other anti-angiogenic therapy. Central Nervous system hemorrhage
Groups:
- Bevacizumab / Irinotecan (Camptosar®, CPT-11): CPT-11 (Irinotecan, Camptosar) - Patients being treated with an enzyme inducing antiepileptic drug (EIAED) will receive 340 mg/m² IV; others will receive 125 mg/m² IV 90 min on days 1 and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / Irinotecan (Camptosar®, CPT-11) | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine
Started | 3 | 0 | 1 | 0 | 2 | 2
Completed | 3 | 0 | 1 | 0 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab / CPT-11: CPT-11 (Irinotecan, Camptosar) - Patients being treated with an enzyme inducing antiepileptic drug (EIAED) will receive 340 mg/m² IV; others will receive 125 mg/m² IV 90 min on days 1 and 15, in combination with avastin 10 mg/kg on days 1 and 15 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / CPT-11 | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine | Total
Number analyzed (Participants) | 3 | 0 | 1 | 0 | 2 | 2 | 8
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0 |  | 0 | 0 | 0
  Between 18 and 65 years | 3 |  | 1 |  | 2 | 2 | 8
  >=65 years | 0 |  | 0 |  | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (NA) — The study did not meet expected accrual |  | 42 (NA) — The study did not meet expected accrual |  | 52.5 (NA) — The study did not meet expected accrual | 56.5 (NA) — The study did not meet expected accrual | 50.6 (5.8)
Gender [Number; unit: participants]
  Female | 3 |  | 1 |  | 2 | 2 | 8
  Male | 0 |  | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 1 |  | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Will be Assessed According to Standard (CTCAE Version 3.0) Toxicity Reporting Criteria.
Description: Primary endpoint has not been analysed secondary to slow and low accrual numbers.
Time Frame: May 2009
Population: Endpoint has not been analysed secondary to slow and low accrual numbers.
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / CPT-11 | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Assess the Activity of Avastin When Added to Single Agent Chemotherapy, as Measured by Radiographic Response Rate,Progression Free Survival, and Overall Survival.
Description: Due to slow accrual study was prematurely closed and endpoint not analysed
Time Frame: 8 to 9 weeks
Population: Due to slow accrual study was prematurely closed and endpoint not analysed
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / CPT-11 | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Determining the Safety and Tolerability of Adding Avastin to Single Agent Chemotherapy to Treat Patients With Brain Metastasis Originating From Breast Cancer
Description: Due to slow accrual study was prematurely closed and endpoint not analysed
Time Frame: trial closure
Population: Due to slow accrual study was prematurely closed and endpoint not analysed
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / CPT-11 | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: To Assess the Quality of Life During Treatment With This Therapeutic Approach
Description: Due to slow accrual study was prematurely closed and endpoint not analysed
Time Frame: 8 to 9 weeks
Arm/Group | Bevacizumab / Capecitabine | Bevacizumab / Docetaxel | Bevacizumab / CPT-11 | Bevacizumab / Paclitaxel | Bevacizumab /Vinorelbine Tartrate | Bevacizumab / Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Avastin (Bevacizumab)/ Capecitabine (Xeloda) | Avastin (Bevacizumab) / Camptosar (CPT 11/ Irinotecan) | Avastin (Bevacizumab)/Gemzar(Gemcitabine,Difluorodeoxycytidine | Avastin (Bevacizumab)/Navelbine (Vinorelbine Tartrate)
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/1 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin (Bevacizumab)/ Capecitabine (Xeloda) (N=3) | Avastin (Bevacizumab) / Camptosar (CPT 11/ Irinotecan) (N=1) | Avastin (Bevacizumab)/Gemzar(Gemcitabine,Difluorodeoxycytidine (N=2) | Avastin (Bevacizumab)/Navelbine (Vinorelbine Tartrate) (N=2)
dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 — grade 3, Xeloda/Avastin arm
renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
hypophophatemia (Investigations) | 0 | 0 | 1 | 0
hypokalemia (Investigations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Avastin (Bevacizumab)/ Capecitabine (Xeloda) (N=3) | Avastin (Bevacizumab) / Camptosar (CPT 11/ Irinotecan) (N=1) | Avastin (Bevacizumab)/Gemzar(Gemcitabine,Difluorodeoxycytidine (N=2) | Avastin (Bevacizumab)/Navelbine (Vinorelbine Tartrate) (N=2)
ALT: increased (Hepatobiliary disorders) | 0 | 1 | 0 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
anorexia (General disorders) | 2 | 1 | 1 | 0
AST: elevated (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 1 | 0
Calcium: elevated (Investigations) | 1 | 0 | 0 | 0
heart flutter (Cardiac disorders) | 0 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0
mouth tenderness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Creatinine:elevated (Investigations) | 0 | 1 | 0 | 0
dehydration (General disorders) | 1 | 0 | 0 | 0
dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
edema: limb (General disorders) | 1 | 0 | 1 | 1
fatigue (General disorders) | 3 | 1 | 1 | 2
Flushing (General disorders) | 0 | 1 | 0 | 0
hair loss (General disorders) | 0 | 1 | 0 | 0
heart burn (Gastrointestinal disorders) | 0 | 0 | 0 | 1
hemaglobin (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
nose bleeds (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
hot flashes (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Insomnia (General disorders) | 2 | 1 | 1 | 0
leukocytes (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
libido (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
memory impairment (Psychiatric disorders) | 2 | 1 | 0 | 0
hypokalemia (Investigations) | 1 | 1 | 1 | 1
irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
depression (Psychiatric disorders) | 1 | 0 | 1 | 0
stomatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 0
neuropathy sensory (Nervous system disorders) | 2 | 1 | 0 | 0
neutrophils (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
peripheral vision changes (Eye disorders) | 1 | 1 | 0 | 0
blindness (Eye disorders) | 1 | 0 | 0 | 0
Pain: shingles (General disorders) | 1 | 0 | 0 | 0
Pain: Shoulder and back (General disorders) | 2 | 1 | 1 | 0
Pain: breast (General disorders) | 1 | 0 | 0 | 1
Pain: extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
headache (Nervous system disorders) | 1 | 0 | 1/1 | 1
blurred vision (Eye disorders) | 1 | 0 | 0 | 0
visual floaters (Eye disorders) | 0 | 0 | 0 | 1
voice changes (General disorders) | 0 | 0 | 1 | 1
vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0
weight gain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
joint pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
phosphorus low (Investigations) | 0 | 0 | 1 | 0
sore throat (General disorders) | 1 | 0 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
hand foot syndrome (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
chills/rigors (General disorders) | 1 | 0 | 0 | 1
seizure (Nervous system disorders) | 0 | 0 | 1 | 0
skin breakdown (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
taste changes (Gastrointestinal disorders) | 1 | 0 | 0 | 0
cerebral thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
DVT (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
tremors (Nervous system disorders) | 0 | 0 | 0 | 1
BUN elevated (Investigations) | 0 | 1 | 0 | 0
vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
weight loss (General disorders) | 1 | 1 | 0 | 0
dry mouth (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No